CLINICAL TRIAL: NCT03408418
Title: Tomographic and Histological Evaluation of Postextraction Sockets Treated With Leucocyte- and Platelet-rich Fibrin: a Randomized Clinical Trial
Brief Title: L-PRF in Alveolar Ridge Preservation
Acronym: L-PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, João Vitor dos Santos Canellas, DDS MS, PhD Student, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 72596717.3.0000.5259
Record Dates: First submitted 2018-01-16; First posted 2018-01-24 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Bone Loss, Alveolar
Keywords: Platelet-rich fibrin; Tooth Extraction; Alveolar Bone Grafting
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-PRF group (Experimental): The use of autologous leucocyte- and platelet-rich fibrin in alveolar sockets after dental extraction.
  Interventions: Procedure: Platelet-rich fibrin
- Control (No Intervention): Conventional tooth extraction without any bone substitute.

INTERVENTIONS:
Procedure: Platelet-rich fibrin — The use of autologous platelet-rich fibrin after tooth extraction to promote bone healing and alveolar ridge preservation
  Other Names: platelet concentrate
  Arms: L-PRF group

SUMMARY:
The effect of leucocyte- and platelet-rich fibrin (L-PRF) for enhancing the healing after dental extractions is still a matter of debate. The available literature suggests that L-PRF performs positive effect to improve alveolar preservation resulting in less bone resorption on extraction sockets. L-PRF is a second generation of platelet concentrate produced without biochemical blood manipulation. L-PRF is composed by three key parameters: first, the presence of platelets; second, the presence of leucocytes; third, the density and complex organization of the fibrin matrix architecture produced by a natural polymerization process. The theory is that this key parameters acts to produce a faster bone healing.

ELIGIBILITY:
Inclusion Criteria:

* (1) Health patients, American Society of Anesthesiologists (ASA) I or II
* (2) Patients who need to submit tooth extraction (pre-molar, canine and incisor teeth - uniradicular teeth or teeth with fused roots) which present ideal conditions to receive dental implants after 3 months.

Exclusion Criteria:

* Smoking
* Systemic diseases related with healing disorders
* Poor oral hygiene
* Pregnant or lactating patient
* Use of flap elevation for dental extraction

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Width resorption 1mm | After 3 months
  The ridge width differences between baseline and after three months of healing 1 mm below the crest.

SECONDARY OUTCOMES:
Width resorption 3mm | After 3 months
  The ridge width differences between baseline and after three months of healing 3 mm below the crest.
Width resorption 5mm | After 3 months
  The ridge width differences between baseline and after three months of healing 5 mm below the crest.
Histological Analysis - fibrous tissue | After 3 months
  The percentage of soft (fibrous) tissue
Histological Analysis - bone cells | After 3 months
  Quantity of bone cells (osteoblast, osteoclast and osteocyte)
Histological Analysis - capillary vessels | After 3 months
  Quantity of capillary vessels
Histological Analysis - new bone formation | After 3 months
  The percentage of the newly formed bone

CONTACTS AND LOCATIONS:
Overall Officials: João Canellas, MSc, Principal Investigator — Rio de Janeiro State University
Locations (1):
- Rio de Janeiro State University, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Canellas JVDS, da Costa RC, Breves RC, de Oliveira GP, Figueredo CMDS, Fischer RG, Thole AA, Medeiros PJD, Ritto FG. Tomographic and histomorphometric evaluation of socket healing after tooth extraction using leukocyte- and platelet-rich fibrin: A randomized, single-blind, controlled clinical trial. J Craniomaxillofac Surg. 2020 Jan;48(1):24-32. doi: 10.1016/j.jcms.2019.11.006. Epub 2019 Nov 29. PMID 31810848